CLINICAL TRIAL: NCT01153425
Title: NMR Imaging and Stereological Analysis of Trabecular Bone in Female Subjects 60 and Older at Risk of Fracture Receiving Either Zoledronic Acid or Teriparatide
Brief Title: µMRI of Therapeutic Intervention in Postmenopausal Osteoporosis
Acronym: TERIZOL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Eli Lilly and Company (Industry); Novartis Pharmaceuticals (Industry); National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 803763; R01AR041443 (NIH)
Record Dates: First submitted 2009-06-01; First posted 2010-06-30 (Estimated); Results first posted 2017-08-04 (Actual); Last update posted 2017-08-04 (Actual); Status verified 2017-08

CONDITIONS: Osteoporosis, Osteopenia
Keywords: Osteoporosis; Osteopenia; Fracture Risk; teriparatide or Forteo; zoledronic acid or Reclast
MeSH Terms: conditions — Osteoporosis; Bone Diseases, Metabolic | interventions — Teriparatide; Zoledronic Acid

STUDY DESIGN:
Intervention Model Description: Postmenopausal women, ages ≥ 60 years, indicated for treatment with antiresorptive or anabolic drugs due to severe osteoporosis and high risk of fracture.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Teriparatide (Forteo) (Active Comparator): 20 µg of Teriparatide will be self-injected subcutaneously once a day for 12 months and an MRI at 3T ('Virtual Bone Biopsy') will be performed at 0 and 12 months.
  Interventions: Other: Virtual Bone Biopsy; Drug: Teriparatide
- Zoledronic Acid (Reclast) (Active Comparator): 5 mg of zoledronic Acid will be administered intravenously at baseline and 12 months and an MRI at 3T ('Virtual Bone Biopsy) will be performed at 0 and 12 months.
  Interventions: Other: Virtual Bone Biopsy; Drug: Zoledronic Acid

INTERVENTIONS:
Other: Virtual Bone Biopsy — MRI technology allowing generation of 3D images with considerably smaller voxel size than previous technology through the use of novel pulse sequences and advanced interpolation techniques.
  Other Names: VBB
Drug: Teriparatide — Participants are clinically indicated for treatment.
  Other Names: Forteo
  Arms: Teriparatide (Forteo)
Drug: Zoledronic Acid — Participants are clinically indicated for treatment.
  Other Names: Reclast
  Arms: Zoledronic Acid (Reclast)

SUMMARY:
The purpose of this study is to apply a novel advanced magnetic resonance imaging methodology to evaluate the response to drug intervention involving two treatment arms of postmenopausal participants with osteoporosis, randomized into either a teriparatide (Forteo™) or zoledronic acid (Reclast™) group.

DETAILED DESCRIPTION:
The overall design is to determine and compare the effect of teriparatide and of zoledronic acid on trabecular architecture by magnetic resonance imaging of the midshaft tibia. Post-menopausal women, aged 60 or older with osteoporosis and/or at increased risk of fracture, will be randomized to receive either teriparatide or zoledronic acid. Trabecular microarchitecture, biomechanical parameters and bone mineral density will be examined at 0 and 12 months at 3T MRI.

ELIGIBILITY:
Inclusion Criteria:

* Women
* Age ≥ 60 years
* Bone mineral density T-score of either the spine (L1-L4), total hip or femoral neck of ≤ - 2.0, or has a history of an osteoporotic fracture

Exclusion Criteria:

* Previous treatment with pamidronate, ibandronate, of more than 2 doses in 2 years and of zoledronic acid at any time
* Previous treatment with teriparatide, alendronate or risedronate of more than 2 months in the last 24 months
* Previous treatment with calcitonin within the previous year; previous treatment with an estrogen or selective estrogen modulator will not exclude a potential subject unless she has been taking it for < 1 year (a woman who discontinued estrogen or a selective estrogen receptor within the previous year will also be excluded)
* Other diseases known to affect bone, such as Paget's disease, Cushing's disease, hyperthyroidism, hyperparathyroidism, bone cancer and metastases to bone, and vitamin D deficiency
* Medications known to affect bone, such as anticonvulsants, high dose glucocorticoids (20 mg/day or more > 2 weeks within the previous 6 months)
* Current alcohol use > 3 drinks/day
* Untreated or unstable cardiac, pulmonary, liver (SGOT > 2X upper limit of normal) or renal disease (creatinine > 1.2 mg/dL) or uncontrolled diabetes (hemoglobin A1C > 8.0)
* Prior radiation therapy to the skeleton
* Cardiac pacemakers, ferromagnetic implants or brain aneurysm clips
* Claustrophobia
* Subjects whose initial MRI is of poor quality due to motion artifact will be asked to repeat the examination; if a repeat MRI is of poor quality due to motion artifact, the subject will be excluded from the study
* Abnormalities of the which delay esophageal emptying such as stricture or achalasia
* Inability to stand or sit upright for at least 30 minutes
* Hypocalcemia
* Uric acid level >7.5ml/dl
* Subjects with metallic objects in their bodies

Min Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Postmenopausal women
Enrollment: 33 (Actual)
Dates: Start 2008-07; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Felix W. Wehrli, Ph.D., Principal Investigator — University of Pennsylvania, Department of Radiology; Peter J. Snyder, M.D., Study Director — University Of Pennsylvania, Department of Endocrinology
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the Philadelphia region via various modes of public advertisements (radio, newspapers, flyers).
Pre-assignment Details: To qualify for participation participants must have BMD T-scores of either the spine (L1-L4) or total hip of ≤ -2.5 or a history of osteoporotic fracture.
Groups:
- Teriparatide (Forteo): 20 µg of Teriparatide will be self-injected subcutaneously once a day for 24 months and an MRI ('Virtual Bone Biopsy') will be performed at 0 and 24 months.
  Virtual Bone Biopsy by Magnetic Resonance Imaging: The MRI involves virtual bone biopsy technology currently being developed. This new technology is not commercially or elsewhere available. It allows generation of 3D images of considerably smaller voxel size than the previous technology by employing new pulse sequences and advanced interpolation techniques. The enhanced resolution will enable capturing subtle remodeling-induced changes, such as reversal of the fenestration caused by prior osteoclastic resorption cavities. It will also permit measurement of trabecular thickness with increased accuracy and precision. Advances have also been made toward superior registration of follow-up scans relative to the baseline scans. This, we project, provides improved reproducibility and thus increased statistical power.
- Zoledronic Acid (Reclast): 5 mg of zoledronic Acid will be administered intravenously at baseline and 12 months and an MRI ('Virtual Bone Biopsy) will be performed at 0 and 24 months.
  Virtual Bone Biopsy by Magnetic Resonance Imaging: The MRI involves virtual bone biopsy technology currently being developed. This new technology is not commercially or elsewhere available. It allows generation of 3D images of considerably smaller voxel size than the previous technology by employing new pulse sequences and advanced interpolation techniques. The enhanced resolution will enable capturing subtle remodeling-induced changes, such as reversal of the fenestration caused by prior osteoclastic resorption cavities. It will also permit measurement of trabecular thickness with increased accuracy and precision. Advances have also been made toward superior registration of follow-up scans relative to the baseline scans. This, we project, provides improved reproducibility and thus increased statistical power.
Period: Overall Study
Arm/Group | Teriparatide (Forteo) | Zoledronic Acid (Reclast)
Started | 16 | 17
Completed | 13 | 14
Not Completed | 3 | 3
Not completed — Withdrawal by Subject | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Teriparatide (Forteo) | Zoledronic Acid (Reclast) | Total
Number analyzed (Participants) | 16 | 17 | 33
Age, Continuous [Mean (Full Range); unit: years] | 69.55 [58 to 84] | 66.22 [58 to 84] | 67.94 [58 to 84]
Sex: Female, Male [Count of Participants; unit: Participants] — Post menopausal females
  Participants
    Female | 16 | 17 | 33
    Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 16 | 17 | 33
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 12 | 12 | 24
  More than one race | 4 | 5 | 9
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Change in Trabecular Surface-to-curve Ratio
Description: Ratio of the volume densities of surface (S) and curve (C)-type voxels, S/C
Time Frame: Change between baseline and 12 months
Population: Mean change in structural and mechanical markers of bone turnover between the two groups.
Measure: Mean (Standard Deviation); unit: Percentage of Change
Groups:
- Teriparatide (Forteo): 20 µg of Teriparatide self-injected subcutaneously once a day for 24 months with MRI performed at 0, 12 and 24 months.
  The data showed strong increases in finite element derived axial stiffness and improvement in structural parameters indicative of a more connected, more plate-like topology at the 12 and 24-month time points: bone marrow density (BMD), bone volume fraction (BVF), the topological parameters surface-to-curve ratio (S/C), which is a measure of the bone's "platelikeness", erosion index (EI), a parameter expressing the loss of connectivity, and axial stiffness (Ezz), all changed in the direction suggesting an improvement of bone quality.
  No difference was detected between the two treatment arms.
- Zoledronic Acid (Reclast): 5 mg of zoledronic Acid administered intravenously at baseline and 12 months and MRI performed at 0, 12, and 24 months.
  The data showed strong increases in finite element derived axial stiffness and improvement in structural parameters indicative of a more connected, more plate-like topology at the 12 and 24-month time points: bone marrow density (BMD), bone volume fraction (BVF), the topological parameters surface-to-curve ratio (S/C), which is a measure of the bone's "platelikeness", erosion index (EI), a parameter expressing the loss of connectivity, and axial stiffness (Ezz), all changed in the direction suggesting an improvement of bone quality.
  No difference was detected between the two treatment arms.
Arm/Group | Teriparatide (Forteo) | Zoledronic Acid (Reclast)
Number analyzed (Participants) | 13 | 14
Percentage of Change | 9.1 (2.0) | 7.1 (2.6)

2. Secondary Outcome: Percentage of Change in Bone Volume Fraction (BVF)
Description: Average fractional content of bone expressed in percent
Time Frame: Change between baseline and 12 months
Measure: Mean (Standard Deviation); unit: Percentage of Change
Groups:
- Teriparatide (Forteo): 20 µg of Teriparatide self-injected subcutaneously once a day for 24 months with MRI performed at 0 and 24 months.
  The data showed strong increases in finite element derived axial stiffness and improvement in structural parameters indicative of a more connected, more plate-like topology at the 12 and 24-month time points: bone marrow density (BMD), bone volume fraction (BVF), the topological parameters surface-to-curve ratio (S/C), which is a measure of the bone's "platelikeness", erosion index (EI), a parameter expressing the loss of connectivity, and axial stiffness (Ezz), all changed in the direction suggesting an improvement of bone quality.
  No difference was detected between the two treatment arms.
Arm/Group | Teriparatide (Forteo) | Zoledronic Acid (Reclast)
Number analyzed (Participants) | 13 | 14
Percentage of Change | 1.0 (0.8) | 0.6 (0.3)
Statistical Analysis 1: Comparison: Teriparatide (Forteo) vs Zoledronic Acid (Reclast); paired t-test for change from baseline to 24 months; Test type: Other — unpaired t-test for the difference of the means between the two arms; p > 0.05, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 2 years
Description: Adverse events were monitored/assessed without regard to the specific adverse event term. Please note that adverse events do include abnormal laboratory values at screening.
Groups:
- Teriparatide (Forteo): 20 µg of teriparatide will be self-injected subcutaneously once a day for 24 months and an MRI ('Virtual Bone Biopsy') will be performed at 0 and 24 months.
  Virtual Bone Biopsy: MRI technology allowing generation of 3D images with considerably smaller voxel size than previous technology through the use of novel pulse sequences and advanced interpolation techniques.
  Teriparatide: Participants are clinically indicated for treatment.
- Zoledronic Acid (Reclast): 5 mg of zoledronic Acid will be administered intravenously at baseline and 12 months and an MRI ('Virtual Bone Biopsy) will be performed at 0 and 24 months.
  Virtual Bone Biopsy: MRI technology allowing generation of 3D images with considerably smaller voxel size than previous technology through the use of novel pulse sequences and advanced interpolation techniques.
  Zoledronic Acid: Participants are clinically indicated for treatment.
Arm/Group | Teriparatide (Forteo) | Zoledronic Acid (Reclast)
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/17
Serious Adverse Events (participants affected / at risk) | 1/16 | 0/17
Other Adverse Events (participants affected / at risk) | 15/16 | 12/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Teriparatide (Forteo) (N=16) | Zoledronic Acid (Reclast) (N=17)
Serious (Surgical and medical procedures) | 1 (1) | 0 (0) — Surgical intervention for meningioma
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Teriparatide (Forteo) (N=16) | Zoledronic Acid (Reclast) (N=17)
Moderate (Gastrointestinal disorders) | 0 (0) | 1 (1)
Moderate (General disorders) | 0 (0) | 2 (2)
Moderate (Blood and lymphatic system disorders) | 2 (3) | 0 (0) — Hypercalcemia
Moderate (Eye disorders) | 1 (1) | 0 (0) — Beginning of detached retina
Moderate (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Abrasions from fall
Moderate (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Dog bite
Moderate (Surgical and medical procedures) | 0 (0) | 1 (1) — Extractions due to dental disease
Moderate (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Edema of finger
Moderate (Surgical and medical procedures) | 1 (1) | 0 (0) — Surgical repair of uterine prolapse
Mild (Blood and lymphatic system disorders) | 7 (9) | 6 (12) — Abnormal lab values
Mild (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) — Sinus Infection
Mild (General disorders) | 9 (11) | 4 (4) — Non-Specific
Mild (Eye disorders) | 0 (0) | 1 (1) — Eye Redness

LIMITATIONS AND CAVEATS:
Insufficient Power

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No